CLINICAL TRIAL: NCT04289220
Title: A Phase I Clinical Trial of Anti-CD19 Chimeric Antigen Receptor in PiggyBac Transposon-Engineered T Cells for the Treatment of Patients With Relapsed/Refractory/High-risk B-cell Lymphoma or B-cell Acute Lymphoblastic Leukemia
Brief Title: Anti-CD19 CAR in PiggyBac Transposon-Engineered T Cells for Relapsed/Refractory B-cell Lymphoma or B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1-N-25318000002027
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: B Cell Lymphoma; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 CAR-T Cells Injection (Experimental): Anti-CD19 CAR-T Cells Injection, Dosage form：injection Dosage:1-2.5x10^6/kg, 100ml/time, The CAR-T cells will be administered by i.v. injection over 20-30 minutes, Frequency: total one time
  Interventions: Biological: Anti-CD19 CAR-T Cells Injection

INTERVENTIONS:
Biological: Anti-CD19 CAR-T Cells Injection — Dosage form：injection Dosage:1-2.5x10^6 cells/kg, 100ml/time, The CAR-T cells will be administered by i.v. injection over 20-30 minutes, Frequency: total one time

SUMMARY:
Our previous study demonstrated that anti-CD19 chimeric antigen receptor in piggyBac transposon-engineered T cells have strong tumor-killing activity in vitro and therapeutic effects in cell line-derived xenograft models, and no obvious side effects such as neurotoxicity and cytokine storm occurred. Therefore, we want to evaluate the safety and clinical effect of anti-CD19 CAR-T cells in clinical trials.

DETAILED DESCRIPTION:
Using piggyBac transposon/transposase system to deliver genes into primary human T cells - example expression of CD19 CAR.CARs specific to the human CD19 antigen were used. All CARs contained the scFv against human CD19 (clone FMC-63), The third BBz CD28z CAR consisted of the scFv linked to the intracellular domains of CD28, 4-1BB and CD3z through a CD28 transmembrane domain;

Subjects with relapsed/refractory CD19-positive B-cell Lymphoma or B-ALL can participate if all eligibility criteria are met. All patients received chemotherapy with fludarabine and cyclophosphamide before the infusion of anti-CD19 CAR-T cells.. After the infusion, subjects will accept follow-up for side effects and effect of anti-CD19 CAR-T cells.

Follow-up :

Safety and adverse events (safety and tolerability of anti-CD19 CAR-T cell therapy within 14 days): The number and severity of adverse events, an evaluation of their association with the anti-CD19 CAR-T cell treatment, and the outcome of the adverse events. Possible adverse events include cytokine release syndrome, hypotension, reversible neurotoxicity, hypogammaglobulinemia, etc. CT was used to evaluate B-lymphoma lesions. B-ALL bone marrow samples were collected by bone marrow aspiration to assess minimal residual disease. Flow cytometry was used to detect proportion of T cells, B cells, and NK cells in the blood, and expression of CD3, CD4, CD8, anti-CD19 CAR to determine the effect of anti-CD19 CAR-T treatment. Plasma levels of the cytokines IFN-gamma, TNF-α, IL-2, GM-CSF, IL-10, and IL-6 were also determined.

Data analysis:

Overall survival and progress free survival were determined by the Kaplan-Meier method, using all enrolled patients to determine overall survival.

Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the Informed Consent Document;
2. Male or female patients aged 18 to 70 years (inclusive);
3. Pathologically and histologically confirmed CD19 + B cell tumors; Patients currently have no effective treatment options, such as chemotherapy or relapse after hematopoietic stem cell transplantation; Or patients voluntarily choose transfusion of anti-CD19 CAR-T cells as the first treatment program;
4. B-cell tumors / lymphomas and B-cell acute lymphoblastic leukemia include the following four types:1) B-cell acute lymphoblastic leukemia;2) Indolent B-cell lymphomas;3) Aggressive B-cell lymphoma; 4) Multiple myeloma;
5. Subjects:

(1) Residual lesions remain after treatment and Not suitable for Hematopoietic stem cell transplantation (auto/allo-HSCT); (2) Relapse after Complement receptor 1 (CR1) and unsuitable for HSCT; (3) Patients with high risk factors; (4) Relapse or no remission after hematopoietic stem cell transplantation or cell immunotherapy.

6. Have measurable or evaluable tumor foci;

7. Liver, kidney and cardiopulmonary functions meet the following requirements:

1) Serum glutamic pyruvic transaminase (ALT) and serum glutamic oxaloacetic transaminase (AST) <3 ×upper limit of normal (ULN);2) Total bilirubin ≤34.2μmol/L;3) Serum creatinine<220μmol/L;4) Baseline oxygen saturation≥95%;5) Left ventricular ejection fraction（LVEF）≥40%.

8. Subjects who did not receive Chemotherapy, Radiotherapy, Immunotherapy (immunosuppressive drugs) or other treatment within 4 weeks prior to enrollment; Relevant toxicity≤1 grade before enrollment (except for low toxicity such as hair loss);

9. Peripheral superficial venous blood flow is smooth, which can meet the needs of intravenous drip;

10. Clinical performance status of eastern cancer cooperation group (ECOG) score ≤2,Expected survival≥3 months;

Exclusion Criteria:

1. Pregnant (urine/blood pregnancy test positive) or lactating women;
2. Planned pregnancy during treatment or within 1 year after treatment, or a male subject whose partner plans pregnancy within 1 year of their cell transfusion;
3. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 year after enrollment;
4. Active or uncontrollable infection within four weeks prior to enrollment;
5. Patients with active hepatitis B/C;
6. HIV-infected patients;
7. Severe autoimmune or immunodeficiency disorders;
8. Patients are allergic to macromolecule drugs such as antigens or cytokines;
9. Subjects participated in other clinical trials within 6 weeks before enrollment;
10. Systematic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Mental illness;
12. Drug abuse/addiction;
13. The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Grade and number of cytokine release syndrome and neurotoxic effects in participants receiving treatment | 14 day
  Anti-CD19 CAR-T cells growing use requires further education/training and prompt management of safety and tolerability.
Persistence of anti-CD19 CAR-T cells in participants | 1 year
  Copies numbers of CAR in peripheral blood (PB)

SECONDARY OUTCOMES:
Overall survival | 3 years
  For all subjects, overall survival refers to the period from being included in the test group to death caused by any reason
Progress Free Survival | 3 years
  Progression-free survival refers to the period between the start of treatment for participants and the observation of disease progression or death for any reason.
Duration of Response after administration | 3 years
  Duration of Response after administration

CONTACTS AND LOCATIONS:
Overall Officials: Zongliu Hou, Study Director — Kunming Yan'an Hospital
Locations (1):
- Kunming Yan'an Hospital, Kunming, Yunnan, China